## THE EFFECT OF THE CHECK LIST DEVELOPED FOR DRUG ADMINISTRATION FROM ENTERAL NUTRITION TUBE ON ADMINISTRATION ERRORS

## 08.02.2022

## INFORMED CONSENT FORM

Dear participant; This research is carried out to examine the effect of the checklist, which is planned to be developed for drug administration from enteral feeding tube, in practice. With the checklist, the validity and reliability of which will be tested, it is expected that the erroneous applications encountered in drug administrations from the enteral feeding tube will decrease. Your participation in this study is entirely voluntary. You have the right to refuse to participate in the research. If you agree to participate in this research, you will first be asked to answer a 16-question questionnaire. Secondly, the researcher will make an observation with the video recording of your enteral drug administration, and then you will be asked to answer another 20 questions on the subject. After the planned checklist has been developed, the observation and the second survey will be repeated. Considering your workload, you are expected to allocate a maximum of 5-10 minutes for work. Your answers to the questions will be kept confidential and will only be evaluated by the researcher and used for this research purpose only. You must answer each question in the questionnaire given to you for the purpose of data collection sincerely and accurately for the research to be reliable. Thank you for your interest and help.

Note: In order for the researcher to participate in your applications, your shift hours must be known. For this purpose, your contact information is needed in order to be able to contact you directly.

Principal Investigator: Emel KÜLEKCİ,

Ph.D. Student of the Department of Surgical Diseases Nursing

Tel: 05062712760

Signature:

Advisor: Prof. Dr. Emine IYIGUN

Health Sciences University Gulhane Nursing Faculty Dean

I have read the above information and under these conditions, of my own free will, without any coercion or pressure;

| ( ) I agree to participate in the research. |
|----------------------------------------------------|
| Name and surname: |
| Phone number: |
| Signature: |
| ( ) I do not agree to participate in the research. |
| Name and surname: |